CLINICAL TRIAL: NCT03674606
Title: An Open-label Randomized-Controlled Trial of Early Screening Test for Pre-eclampsia and Growth Restriction
Brief Title: Trial of Early Screening Test for Pre-eclampsia and Growth Restriction
Acronym: TEST
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University College Dublin (Other)
Collaborators: Perinatal Ireland (Other); National Maternity Hospital, Ireland (Other); Royal College of Surgeons, Ireland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TEST_PILOT_V1; 2013-004241-17 (EudraCT Number); ISRCTN15191778 (Registry Identifier: ISRCTN)
Record Dates: First submitted 2018-07-20; First posted 2018-09-17 (Actual); Last update posted 2018-09-17 (Actual); Status verified 2018-09

CONDITIONS: Pre-Eclampsia; Placenta Diseases; Eclampsia Preeclampsia; Fetal Growth Retardation; Foetal Growth Restriction
Keywords: Pre-eclampsia; Fetal Medicine Foundation; FMF screening; First trimester; Aspirin; Placental disease; nulliparous; LDA; low-dose aspirin; fetal growth restriction; trans-abdominal uterine artery doppler examination
MeSH Terms: conditions — Pre-Eclampsia; Placenta Diseases; Fetal Growth Retardation | interventions — Aspirin

STUDY DESIGN:
Intervention Model Description: Three-armed parallel, multi-center, open-label randomised control trial
Oversight: Data Monitoring Committee: Yes | US Export: Yes

ARMS (3):
- Routine low-dose aspirin (Experimental): Subjects shall receive standard antenatal care as well as taking oral low-dose aspirin from the eligibility visit until 36-week gestation once daily, as prescribed by the research clinician. Fetal Medicine Foundation screening test results from the recruitment visit shall not be disclosed to the participants in this arm.
  Interventions: Drug: Low dose aspirin
- No aspirin (No Intervention): No low-dose aspirin will be prescribed. Fetal Medicine Foundation screening test results from the recruitment visit shall not be disclosed to the participants in this arm.
- Test-indicated low-dose aspirin (Active Comparator): The Fetal Medicine Foundation screening test will be used to determine whether a subject is at high risk of developing any pre-eclampsia until 42-week gestation. Participants with risk > 1:8 must start low-dose aspirin treatment immediately. Participants with a risk < 1:8 will be excluded.
  Interventions: Drug: Low dose aspirin

INTERVENTIONS:
Drug: Low dose aspirin — One 75 mg aspirin dose taken daily
  Other Names: Nu-Seals 75; 75 mg aspirin
  Arms: Routine low-dose aspirin; Test-indicated low-dose aspirin

SUMMARY:
A study of aspirin use in pregnancy to prevent high blood pressure and growth restriction of the fetus

DETAILED DESCRIPTION:
Ischemic placental disease (IPD) is an entity encompassing pre-eclampsia, fetal growth restriction (FGR) and placental abruption and has a combined incidence in pregnancy of 10-15%. Pre-eclampsia is a serious systemic condition affecting 3-5% of pregnancies and is responsible for > 50,000 of maternal deaths annually worldwide. The International Society for the Study of Hypertension in Pregnancy defines pre-eclampsia as gestational hypertension with proteinuria of 300 mg or more in 24 h.

The use of low dose aspirin (LDA) prior to 16-weeks' gestation can prevent the pathological process causing placental disease by altering the balance of prostacyclin and thromboxane; hence preventing spiral artery thrombosis and widespread endothelial dysfunction.

There is extensive evidence, demonstrating the efficacy and safety of LDA for prevention of placental disease in high-risk pregnancies where there are clearly identifiable risk factors. However, there is a paucity of research into its efficacy in low-risk women. Administration of aspirin in pregnancy is associated with absolute risk reductions of 2% to 5% for pre-eclampsia, 1% to 5% for FGR 2% to 4% for preterm delivery with no associated increase in perinatal or maternal morbidity.

Several screening tests have been devised to detect the risk of pre-eclampsia and FGR from the first trimester. One of the most notable is that of The Fetal Medicine Foundation (FMF), UK that have devised an algorithm encompassing uterine artery Doppler pulsatility indices, mean arterial pressure (MAP), the placental biomarkers PAPP-A and PLGF in addition to maternal characteristics, which can detect 96% of cases of pre-eclampsia requiring delivery before 34 weeks and 54% of all cases of pre-eclampsia at a fixed false-positive rate of 10%. The FMF screening test is reserved as a research tool, pending validation within a low-risk population. Thus far it has been externally validated in other studies of unselected women with conflicting results as to sensitivity and specificity for placental disease prediction. Following validation of the FMF screening test in low-risk nulliparous women, which is currently the topic of on-going research, the FMF pre-eclampsia screening test may potentially come into clinical practice in the future. Current guidelines followed within the UK, set by The National Institute for Health and Clinical Excellence advocate screening through history taking and provision of LDA in the presence of one major risk factor or two moderate risk-factors. The American College of Obstetricians and Gynecologists have a similar stance and do not recommend screening to predict pre-eclampsia beyond obtaining an appropriate medical history to evaluate for risk factors. They recommend that any further screening tests beyond this should undergo a cost-effectiveness analysis before being used in routine practice.

It has been postulated that it is more cost-effective to use prophylactic medication, notably aspirin for the prevention of placental disease rather than screening and treating an entire low-risk population. The reason for this is because aspirin is felt to be an effective, affordable and safe treatment in pregnancy.

In light of such evidence, with an emerging novel screening test for pre-eclampsia and the efficacy of LDA for placental disease prevention it may be more clinically effective and affordable to prescribe LDA routinely to all women in their first pregnancy as opposed to being upon the basis of a screening test. To assess this hypothesis a preliminary pilot study is required to determine feasibility, acceptability and statistical power required for such a study. The study proposed is a three-armed parallel, multi-center, open-label randomized control trial (RCT) in low-risk women to determine; (i) the efficacy and (ii) the acceptability of women to take routine LDA, versus no LDA versus LDA on the basis of a pre-eclampsia screening test in their first pregnancy. It can be anticipated that the use of such a three-armed study will aid in determining if it is more acceptable to women and feasible to prescribe LDA routinely compared to not at all, or based on results of a screening test.

ELIGIBILITY:
Inclusion Criteria:

* Nulliparous women.
* Ability to speak and .read English
* Singleton pregnancy at <14 weeks.
* Willing to sign voluntarily a statement of informed consent to participate in the study.

Exclusion Criteria:

* Presence of fetal anomaly at the time of the first trimester scan
* Women with known major risk factors for pre-eclampsia who should already be on Aspirin as per National Institute of Clinical Excellence (NICE) guidance; specifically chronic hypertension, underlying connective tissue, renal or vascular disorder, type 1 diabetes mellitus.
* Under 18 years of age.
* Currently enrolled in other clinical trials.
* Contraindications to Aspirin therapy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Eligibility will be assessed based on first pregnancy status.
Enrollment: 546 (Actual)
Dates: Start 2014-02-01 (Actual); Primary Completion 2016-04-13 (Actual); Study Completion 2016-04-13 (Actual)

PRIMARY OUTCOMES:
The proportion of eligible women that agree to participate in the study | Throughout study completion, less than 40 weeks
  The proportion of eligible women that agree to participate in the study - this will be reflected as a proportion of the number of women approached at the screening stage (feasibility)
Adherence to aspirin if prescribed | 36 weeks
  Rate of adherence among study subjects prescribed aspirin.
The proportion of study subjects in whom it is possible to obtain first trimester trans-abdominal uterine artery Doppler examination | 36 weeks
  This outcome includes the subjectively recorded ease of acquisition (feasibility).
The proportion of study subjects with a completed screening test who are issued the screening result within one week of having the test performed | 1 week
  This includes the number of women within the screen and treatment group that went beyond 16-weeks before receiving the screening test result as beyond this time LDA may not be effective (feasibility).
Attendance at study visits | 36 weeks
  Rate of attendance of study visits by study subjects
Satisfactory collection of all endpoints and variables | 36 weeks
  Proportion of study subjects on which data for all other endpoints can be collected
Any specific study protocol violations | 36 weeks
  Proportion of study subjects for which protocol violations are recorded

SECONDARY OUTCOMES:
The rate of pre-eclampsia as defined by the International Society for the Study of Pre-eclampsia in Pregnancy. | Childbirth
The rate of fetal growth restriction. | Childbirth
Spontaneous or iatrogenic delivery. | Prior to 34 and 37 completed weeks of gestation
Rate of admission to the neonatal intensive care unit. | Childbirth
  rate of placental abruption, any reported death (stillbirth, neonatal or infant death) and small for gestational age infants.
Patient acceptability: ease of swallowing medication proportioned between categories of a 5-point Likert scale from "strongly agree" to "strongly disagree" | 20--22 weeks
  Proportion of subjects who either 1) "strongly agree", 2) "agree", 3) neither agree/disagree", 4) disagree or 5) strongly disagree with the statement "Aspirin was easy to swallow".
Patient acceptability: reasons of failing compliance with study intervention regimen proportioned between answers to a 5-point multiple-choice question. | 20--22 weeks
  Proportion of subjects who chose either "Reservations of taking aspirin", "Bleeding", "It caused stomach upset", "I forgot" or "Other" as a reason for missing aspirin dose.
Patient acceptability: opinions on the screening test proportioned between categories of a 3-point rating scale ranging from "Useful" to "Inconvenient" | 20--22 weeks
  Proportion of subjects who chose either 1) "Useful", 2) "Neither useful/inconvenient" or 3) "Inconvenient" to complete the statement "With regards the screening test I found it"
Patient acceptability: opinions for taking study intervention in the future proportioned between answers to a 3-point multiple-choice question. | 20--22 weeks
  Proportion of subjects who chose either "Take aspirin routinely", "Take aspirin only if I was at risk" or "Neither" to complete the statement "In a future pregnancy I would"

CONTACTS AND LOCATIONS:
Locations (2):
- Ireland (2):
  - National Maternity Hospital, Dublin
  - Rotunda Hospital, Dublin

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Mone F, Mulcahy C, McParland P, Stanton A, Culliton M, Downey P, McCormack D, Tully E, Dicker P, Breathnach F, Malone FD, McAuliffe FM. An open-label randomized-controlled trial of low dose aspirin with an early screening test for pre-eclampsia and growth restriction (TEST): Trial protocol. Contemp Clin Trials. 2016 Jul;49:143-8. doi: 10.1016/j.cct.2016.07.003. Epub 2016 Jul 6. PMID 27394381